CLINICAL TRIAL: NCT05446012
Title: Ectopic Pregnancy and Thyroid Disorders
Brief Title: Relationship Between Ectopic Pregnancy and Thyroid Disorders
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Serif Aksin, associate professor, Siirt University
Other Study IDs: SiirtU
Record Dates: First submitted 2022-06-26; First posted 2022-07-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Ectopic Pregnancy; Thyroid Diseases; Pregnancy, Ectopic
Keywords: Thyroid disorders; pregnancy; Ectopic
MeSH Terms: conditions — Pregnancy, Ectopic; Thyroid Diseases; Choristoma | interventions — Thyroid Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women diagnosed with ectopic pregnancy (n: 40): thyroid function tests (TSH, sT3, sT4, TT3, TT4, thryoglobulin, Anti-Peroxidase Antibody, Anti- thryoglobulin Antibody, TSH receptors antibody levels) will be done in women diagnosed with ectopic pregnancy
  Interventions: Diagnostic Test: thyroid function tests
- Control group pregnants (n:40): thyroid function tests (TSH, sT3, sT4, TT3, TT4, thryoglobulin, Anti-Peroxidase Antibody, Anti- thryoglobulin Antibody, TSH receptors antibody levels) will be done in pregnant women in early pregnancy week.
  Interventions: Diagnostic Test: thyroid function tests

INTERVENTIONS:
Diagnostic Test: thyroid function tests — blood sample for thyroid function tests (TSH,T3,T3,Anti peroxidase antibody, anti thyroglobulin antibody)

SUMMARY:
Fallopian tubes participate in the incorporation of gametes and embryos into the endometrial cavity. It also provides an optimal environment for flattening and early embryonic development. Tubal pathologies can cause both primary and secondary infertility. This condition has been associated with overt and subclinical hypothyroidism. However, the effects of hypothyroidism on tubal activity are not fully known. Although a few animal experiment studies on this subject have been published, there is no study on this subject in the literature. Demonstrating that epithelial and smooth muscle cells of rat fallopian tubes express thyroid receptors in animal experiments showed that fallopian tubes are targets for thyroid hormones. Again, in an animal experiment study, it was revealed that thyroid hormones have an important control on glycogen and lipid storage, lipid signaling and lymphocyte infiltration, which have an important role in maintaining the microenvironment in the rat fallopian tubes. This microenvironment is necessary for fertilization, sperm capacitation and gamete development. In another animal experimental study, it was thought that changes in the size of the epithelium of the fallopian tubes and cell metabolism in hypothyroid rabbits may affect oviductal activity and reproductive functions. An ectopic pregnancy is defined as a pregnancy implanted outside of the uterus. Ectopic pregnancy >98% implants in the fallopian tube. The etiology of ectopic pregnancy is unclear, but tubal implantation is probably due to impaired embryo-tubal transport. This is due to changes in the tubal environment. Based on this information, we aim to determine the possible relationship between hypothyroidism and ectopic pregnancy in humans in our study.

DETAILED DESCRIPTION:
Our aim in this study is to determine the possible relationship between hypothyroidism and ectopic pregnancy in humans. For this purpose, 40 patients with a diagnosis of ectopic pregnancy and 40 patients with diagnosis of early pregnancy followed in Siirt Training and Research Hospital between 30 June 2022 and 30 October 2022 will be included in the study. The patient's age, pregnancy history, medical history and laboratory findings (TSH, sT3, sT4, TT3, TT4, thryoglobulin , Anti-Peroxidase Antibody, Anti-thryoglobulin Antibody, TSH receptors antibody ) will be recorded. In the light of the information gathered, it will be tried to determine whether there is a relationship between thyroid dysfunctions and ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Having an early pregnancy or ectopic pregnancy

Exclusion Criteria:

* using medications due to thyroid gland dysfunction
* history of ectopic pregnancy
* history of tubal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women over 18 years of age diagnosed with ectopic pregnancy or early pregnancy
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Thyroid dysfunction and ectopic pregnancy | Through study completion, an average of 5 months
  TSH, T3, T4, TT3, TT4, Thyroglobulin, Anti peroxidase antibody, Anti thyroglobulin antibody,TSH receptors antibody will be measured in patients diagnosed with ectopic pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, Principal Investigator — Siirt University Medical Faculty Obstetrics and Gynecology Departmant
Locations (1):
- Siirt Üniversity Medical Faculty, Siirt, Turkey (Türkiye)

REFERENCES:
- [Background] Mendez-Tepepa M, Zepeda-Perez D, Espindola-Lozano M, Rodriguez-Castelan J, Arroyo-Helguera O, Pacheco P, Nicolas-Toledo L, Cuevas-Romero E. Hypothyroidism modifies differentially the content of lipids and glycogen, lipid receptors, and intraepithelial lymphocytes among oviductal regions of rabbits. Reprod Biol. 2020 Jun;20(2):247-253. doi: 10.1016/j.repbio.2020.02.004. Epub 2020 Feb 20. PMID 32089504
- [Background] Oner J, Oner H. Immunodetection of thyroid hormone receptor (alpha1/alpha2) in the rat uterus and oviduct. Acta Histochem Cytochem. 2007 Jul 3;40(3):77-81. doi: 10.1267/ahc.06026. PMID 17653299
- [Background] Anaya-Hernandez A, Rodriguez-Castelan J, Nicolas L, Martinez-Gomez M, Jimenez-Estrada I, Castelan F, Cuevas E. Hypothyroidism affects differentially the cell size of epithelial cells among oviductal regions of rabbits. Reprod Domest Anim. 2015 Feb;50(1):104-11. doi: 10.1111/rda.12455. Epub 2014 Nov 18. PMID 25405800